CLINICAL TRIAL: NCT04319939
Title: Diaphragm Ultrasound Measurements With Variations in Modes of Ventilation
Status: Completed | Type: Observational
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Other Study IDs: IRB19-1627
Record Dates: First submitted 2020-01-16; First posted 2020-03-24 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Mechanical Ventilation
Keywords: Diaphragm Ultrasound; Diaphragm Thickness; Control Mode Ventilation; Spontaneous Mode Ventilation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants receiving mechanical ventilation
  Interventions: Other: Assist Control Mode and Pressure Support Mode Mechanical Ventilation

INTERVENTIONS:
Other: Assist Control Mode and Pressure Support Mode Mechanical Ventilation — Diaphragm ultrasound measurements (end expiration and peak inspiration thickness) will be performed in assist control mode and pressure support mode mechanical ventilation in each participant. The participant will thus serve as his/her own control for these interventions.

SUMMARY:
The overall objective of the study is to conduct an observational study involving intensive care unit patients receiving mechanical ventilation and determine if there are differences in diaphragm thickness ultrasound measurements during expiratory and inspiratory phases in a controlled and spontaneous mode. For patients receiving sedatives, an additional set of measurements will be taken during a standard of care interruption of sedatives

DETAILED DESCRIPTION:
In this study diaphragm ultrasound measurements at end-expiration and peak inspiration phases in assist control and pressure support mode in consented patients admitted to the medical intensive care unit. One-time measurements will be obtained during the first 48hrs that the patients are receiving mechanical ventilation. In patients receiving sedatives, additional measurements will be taken after an interruption of sedatives. Measurements will be compared between modes and on assist-control before and after an interruption of sedatives.

Three consecutive images will be obtained by an investigator that is blinded to the mode (controlled vs. spontaneous). Once measurements are obtained, a second investigator will switch to the other mode (controlled vs. spontaneous) and the blinded investigator will obtain three consecutive images after the patient has adjusted to the subsequent mode (one minute). Tidal volumes will be matched between modes as close as possible. The order of modes to ultrasound (controlled then spontaneous or spontaneous then controlled) will be determined by the non-blinded second investigator. Once the ultrasound measurements are obtained by the research team, image acquisition is concluded for the enrolled patient. The ventilator will be programmed back to the original settings determined by the medical ICU team.

The hypothesis is that the end-expiration diaphragm ultrasound measurement will be thicker in spontaneous mode than controlled mode.

ELIGIBILITY:
Inclusion Criteria:

* Patients > 18 years of age
* intubated and mechanically ventilated for < 48 hours at the time of screening

Exclusion Criteria:

* pregnancy
* history of diaphragmatic paralysis
* neuromuscular blockade
* cardiac arrest

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adult patients admitted to the medical intensive care unit and receiving mechanical ventilation
Sampling Method: Probability Sample
Enrollment: 66 (Actual)
Dates: Start 2020-02-05 (Actual); Primary Completion 2022-04-11 (Actual); Study Completion 2022-04-11 (Actual)

PRIMARY OUTCOMES:
End expiratory diaphragm thickness in controlled and spontaneous modes | Less than 48 hours after mechanical ventilation
  Diaphragm ultrasound measurement at end expiration in assist control mode and pressure support mode

SECONDARY OUTCOMES:
Thickening fraction in controlled and spontaneous modes | Less than 48 hours after mechanical ventilation
  Diaphragm ultrasound measurement at end expiration and inspiration to calculate thickening fraction = (peak inspiration thickness - end expiration thickness)/end expiration thickness in assist control and pressure support mode ventilation
Variance in peak inspiration thickness in controlled and spontaneous modes | Less than 48 hours after mechanical ventilation
  Diaphragm ultrasound measurement at peak inspiration in assist control and pressure support
p0.1 measurements in controlled and spontaneous modes | Less than 48 hours after mechanical ventilation
  A measure of respiratory drive obtained from the ventilator in assist control and pressure support

CONTACTS AND LOCATIONS:
Locations (1):
- The University of Chicago Medical Center, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pearson SD, Lin J, Stutz MR, Lecompte-Osorio P, Pohlman AS, Wolfe KS, Hall JB, Kress JP, Patel BK. Immediate Effect of Mechanical Ventilation Mode and Sedative Infusion on Measured Diaphragm Thickness. Ann Am Thorac Soc. 2022 Sep;19(9):1543-1550. doi: 10.1513/AnnalsATS.202111-1280OC. PMID 35404772